CLINICAL TRIAL: NCT04956783
Title: Comparison of the Occurrence of Adverse Effects With Immune Checkpoint Inhibitors Between a Single and Double Dose Regimen
Brief Title: Occurrence of Adverse Effects With Immune Checkpoint Inhibitors Between a Single and Double Dose Regimen
Acronym: ICI DODO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0298
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective evaluation of the impact of a double dose regimen of immunotherapy use in cancer treatment compared to the single-dose regimen on the occurrence of clinically significant adverse events.

The aim of this study is to provide evidence-based arguments to help clinicians to propose the best treatment regimen for each patient.

ELIGIBILITY:
Inclusion criteria:

- Any adult patient with anti-PD-1 or PD-L-1 immune checkpoint inhibitor as monotherapy

Exclusion criteria:

- age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient (over the age of 18) from Montpellier University Hospital or Montpellier Cancer Institute who has initiated an immunotherapy between 01/01/2019 and 31/12/2020 with anti-PD-1 or PD-L-1 immune checkpoint inhibitor as monotherapy (nivolumab, pembrolizumab, atezolizumab, durvalumab, avelumab)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of clinical significant toxicities | 18 months
  To compare the incidence of clinical significant toxicities reported for patients treated with a cancer immunotherapy on a simple dose regiment versus double dose regimen

SECONDARY OUTCOMES:
To describe the incidence | 18 months
  To describe the incidence, type and severity of overall toxicities (serious and non-serious) reported with single and double dose cancer immunotherapy regimens
To identify risk factors for the development of severe toxicity | 18 months
  To identify risk factors for the development of severe toxicity
To describe the management and evolution of toxicities | 18 months
  To describe the management and evolution of toxicities
To describe the clinical oncologic response | 18 months
  To describe the clinical oncologic response

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Maria, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC